CLINICAL TRIAL: NCT03626207
Title: Calibration of Visual Function Evaluation Tests in Patients With Severe Vision Loss
Brief Title: Development of Visual Function Evaluation Method (2)
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: CLR180001
Record Dates: First submitted 2018-08-08; First posted 2018-08-10 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2019-07

CONDITIONS: Retinitis Pigmentosa
Keywords: Retinitis pigmentosa; Visual function evaluation
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retinitis pigmentosa: Retinitis pigmentosa patients with severe visual impairment

SUMMARY:
The objective of this study is to develop the comprehensive visual function evaluation method in severe visually impaired patient.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with severe visual disturbance (count-fingers or worse vision for severe eyes) at the time of obtaining the consent and at screening

Exclusion Criteria:

* Subjects should not have participated in any other clinical trial or clinical study involving visual function evaluation within 6 months
* History of surgery, past history, and complications (cardiac/ hepatic/ renal/ respiratory/ hematological diseases, optic nerve diseases causing marked loss of visual field, and uveitis etc.) that potentially affect evaluation and safety of the study
* Pregnant women
* Subjects who are judged that continuation of the study is difficult during the study period
* Subjects who are employed by the company sponsoring this study, an organization or institution related to this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retinitis pigmentosa
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
Slit-lamp-microscopy | Up to 3 months
  To assess the visual function.
Optical Coherence Tomography (OCT) test | Day 1
  To assess the visual function.
Early Treatment Diabetic Retinopathy Study (ETDRS) | Up to 3 months
  To assess the visual function.
The 25-item National Eye Institute Visual Function Questionnaire (NEI VFQ-25) | Up to 3 months
  NEI VFQ 25 is a questionnaire intended to measure visual function and quality of life. It has 25 questions. The original response of each item are coded as per the NEI VFQ scoring system ranging from 0 (worst) to 100 (best).
The 11-item National Eye Institute Visual Function Questionnaire (NEI VFQ-11) | Up to 3 months
  NEI VFQ 11 is a questionnaire intended to measure visual function and quality of life. It has 11 questions. The original response of each item are coded as per the NEI VFQ scoring system ranging from 0 (worst) to 100 (best).
Nottingham Adjustment Scale Japanese Version (NAS-J) | Up to 3 months
  NAS-J is the Japanese version of NAS which measures psychological adjustment to the visual impairment, and to assess its validity and reliability. The NAS is composed of 7 psychological subscales including anxiety-depression, self-esteem, attitude to disability, locus of control, acceptance of disability, self-efficacy and attributional style. The original response of each item are coded as per the NAS-J scoring system ranging from 0 (lowest psychological adjustment) to 100 (highest psychological adjustment).
Daily living task dependent on vision (DLTV) questionnaire | Up to 3 months
  DLTV is a quality of life questionnaire composed of 22 items to obtain estimates of self-reported ability to perform vision-related tasks in persons with visual impairment. Participants rate items on a four-point scale, with "Can't see to do" (score, 1), "A lot of difficulty" (score, 2), "A little difficulty" (score, 3), and"No difficulty" (score, 4). The original response of each item are coded as per the DLTV scoring system ranging from 0 (worst) to 100 (best).
Table test | Up to 3 months
  To assess the visual function.
Monitor test | Up to 3 months
  To assess the visual function.
Pupillary function test | Up to 3 months
  To assess the visual function.
Full field stimulus threshold testing (FST) | Up to 3 months
  To assess the visual function.
White flash visual evoked potential (VEP) test | Up to 3 months
  To assess the visual function.
Color flash VEP test | Up to 3 months
  To assess the visual function.
Electrically evoked response (EER) test | Up to 3 months
  To assess the visual function.
White flash Electroretinography (ERG) test | Day 1
  To assess the visual function.
Multifocal ERG test | Up to 3 months
  To assess the visual function.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (1):
- Site JP00001, Kobe, Hyōgo, Japan

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.